CLINICAL TRIAL: NCT01850602
Title: A Phase III Study of PA21 in Hemodialysis Patients With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA1301
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2014-11

CONDITIONS: Hemodialysis; Hyperphosphatemia
Keywords: Hemodialysis; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer

ARMS (2):
- PA21 (Experimental)
  Interventions: Drug: PA21
- Sevelamer hydrochloride (Active Comparator)
  Interventions: Drug: Sevelamer hydrochloride

INTERVENTIONS:
Drug: PA21
  Arms: PA21
Drug: Sevelamer hydrochloride
  Arms: Sevelamer hydrochloride

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PA21 in hemodialysis patients with hyperphosphatemia

ELIGIBILITY:
Inclusion Criteria:

* Patients age 20 or older, regardless of gender.
* Receiving stable maintenance hemodialysis 3 times a week.
* Patients not having changed their phosphate binder agent dose, for 4 weeks or more before their observation period start.

Exclusion Criteria:

* Patients having history of a pronounced brain / cardiovascular disorder.
* Patients having severe gastrointestinal disorders.
* Patients having severe hepatic disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- PA21: PA21
- Sevelamer Hydrochloride: Sevelamer hydrochloride
Period: Overall Study
Arm/Group | PA21 | Sevelamer Hydrochloride
Started | 108 | 105
Completed | 94 | 87
Not Completed | 14 | 18
Not completed — Adverse Event | 7 | 10
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Decrease in serum calcium | 2 | 3
Not completed — Increase in serum ferritin | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol Set
Groups:
- Total: Total of all reporting groups
Arm/Group | PA21 | Sevelamer Hydrochloride | Total
Number analyzed (Participants) | 100 | 92 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (11.7) | 60.8 (12.0) | 60.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 39 | 67
  Male | 72 | 53 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 100 | 92 | 192
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Dialysis vintage [Mean (Standard Deviation); unit: months] | 104.9 (79.7) | 102.4 (90.6) | 103.7 (84.8)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean of Serum Phosphorus Concentrations at the End of Treatment
Description: Covariate: Serum phosphorus concentrations at baseline.
Time Frame: 12 weeks
Population: Per Protocol Set
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | PA21 | Sevelamer Hydrochloride
Number analyzed (Participants) | 100 | 92
mg/dL | 5.00 [4.80 to 5.19] | 5.34 [5.13 to 5.55]
Statistical Analysis 1: Comparison: PA21 vs Sevelamer Hydrochloride; Test type: Non-Inferiority — Non-Inferiority margin: 1.0 mg/dL Non-Inferiority was considerd to be confirmed if the upper limit of two-sided confidence interval became 1.0 mg/dL or less; p = 0.020, ANCOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.63 to -0.05]

2. Secondary Outcome: Serum Phosphorus Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21 | Sevelamer Hydrochloride
Number analyzed (Participants) | 100 | 92
mg/dL | 5.01 (1.01) | 5.33 (1.03)

3. Secondary Outcome: Corrected Serum Calcium Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21 | Sevelamer Hydrochloride
Number analyzed (Participants) | 100 | 92
mg/dL | 9.14 (0.68) | 8.91 (0.71)

4. Secondary Outcome: Serum Intact-PTH Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PA21 | Sevelamer Hydrochloride
Number analyzed (Participants) | 100 | 92
pg/mL | 203.6 (117.1) | 253.1 (168.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | PA21 | Sevelamer Hydrochloride
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/105
Serious Adverse Events (participants affected / at risk) | 6/108 | 5/105
Other Adverse Events (participants affected / at risk) | 47/108 | 42/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 (N=108) | Sevelamer Hydrochloride (N=105)
Diverticulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 (N=108) | Sevelamer Hydrochloride (N=105)
Nasopharyngitis (Infections and infestations) | 24 | 24
Constipation (Gastrointestinal disorders) | 2 | 19
Diarrhoea (Gastrointestinal disorders) | 27 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No